CLINICAL TRIAL: NCT02190344
Title: Study to Evaluate the Functionality of an Eight-Channel Paddle Coil System Using MRI
Brief Title: Functionality of an 8-Channel Paddle Coil for Use With MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 019-2014
Record Dates: First submitted 2014-06-16; First posted 2014-07-15 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Prostate in Healthy Males
Keywords: Eight; Channel; Paddle; Coil; MRI; Prostate; Healthy Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functionality of 8-channel paddle coil system (Experimental)
  Interventions: Device: 8-channel paddle coil

INTERVENTIONS:
Device: 8-channel paddle coil — MRI Coil

SUMMARY:
The objective of this study is to determine the functionality of an eight-channel paddle coil system which is to be used in future MRI studies.

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy among men and the second leading cause of cancer death in men. Currently, MRI is the best imaging modality for both detecting prostate cancer and determining the presence of extra-prostatic extension. Multiparametric Magnetic Resonance, combining T2-weighted, diffusion-weighted and dynamic contrast enhanced imaging (DCE-MRI) is recommended as the minimum acceptable standard for prostate MRI examination. However, MPMRI still lacks diagnostic accuracy in the transition zone, where distinguishing cancer from proliferative nodules has proven difficult. DCE-MRI techniques evaluate the time course of signal intensities after administration of a contrast medium and have been used to successfully differentiate benign from malignant tumours, particularly in breast and prostate cancer. Unfortunately, current DCE approaches have high false-positive rates and are limited in distinguishing prostatitis and vascularized BPH nodules from cancer in active surveillance studies. Future studies that employ spectroscopic MR imaging of the prostate after administration of Hyperpolarized (13C) Pyruvate Injection, are expected to provide a robust, non-invasive method to assist in detecting and characterizing prostate cancer. The objective of this study is to determine the functionality of an eight-channel paddle coil system which is to be used in future Hyperpolarized (13C) Pyruvate Injection studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 80 years of age

Exclusion Criteria:

* Any contra-indication for MR imaging (such as pacemakers, surgical implants, foreign metal objects in the body)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Ability of Coil to produce MRI images | 1 hour
  1. functional with adequate SNR
  2. functional with non-adequate SNR
  3. non-functional

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cunningham, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada